CLINICAL TRIAL: NCT01816061
Title: Executive Functioning in TBI From Rehabilitation to Social Reintegration: COMPASS
Acronym: COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: D0637-R
Record Dates: First submitted 2013-03-19; First posted 2013-03-21 (Estimated); Results first posted 2019-09-11 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Traumatic Brain Injury; Post-Traumatic Stress Disorder
Keywords: Veterans Health; Social Adjustment; Traumatic Brain Injury (TBI); Post-Traumatic Stress Disorder (PTSD); Independent Living; Goals; Education
MeSH Terms: conditions — Brain Injuries, Traumatic; Stress Disorders, Post-Traumatic; Social Adjustment

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental - COMPASS (Experimental): Goal-setting sessions
  Interventions: Behavioral: Experimental - COMPASS
- Control - COMPASS (Active Comparator): Informative phone calls
  Interventions: Behavioral: Control - COMPASS

INTERVENTIONS:
Behavioral: Experimental - COMPASS — Controlled randomized clinical trial. Fifty-five participants in the intervention group will receive eight goal self-management sessions over a period of approximately ten weeks.
  Arms: Experimental - COMPASS
Behavioral: Control - COMPASS — Increased hours of patient-provider interactions Group.
  Other Names: Supported discharge group
  Arms: Control - COMPASS

SUMMARY:
Interventional, controlled clinical trial with two arms, 110 Veterans with TBI and PTSD

DETAILED DESCRIPTION:
The COMPASS (Community Participation through Self-Efficacy Skills Development) program aims at developing and testing a novel patient-centered intervention framework that can be utilized as a platform for VA community re-integration comparative effectiveness research. The COMPASSgoal intervention will be developed and implemented to meet these needs. COMPASSgoal will integrate principles and best practices of goal self-management. Goal setting is a core skill in self-management training by which persons with chronic health conditions learn to improve their status and decrease symptom impact.3F One important mechanism of action of this program appears to be its positive effect on self-efficacy, or confidence in one's ability to attain goals and solve problems.4F

The study goal is to gather data on the efficacy of a novel approach to psychosocial rehabilitation for Veterans with executive function impairment due to traumatic brain injury (TBI), and to explore over time, through relevant measures, Veteran responsiveness to intervention. Veterans with mild TBI will be randomized into two groups: the COMPASS (Community Participation through Self-Efficacy Skills Development) goal-management intervention group and the supported discharge group.

110 participants with residual deficits in executive function due to TBI will be recruited at a minimum of 3 months post-injury from the TBI program at the DC VAMC over the three-year period of the study. The operational definition of executive dysfunction/ inclusion into the study is based on both clinical diagnosis by a study physician and a standardized executive dysfunction measure, the Frontal Systems Rating Scale (FrSBe score), such that a total score or any of the 3 subscale scores < 1 SD compared to the normative score would indicate executive dysfunction sufficient to include in the study. The treatment phase for the Veterans enrolled in the intervention group will continue for two consecutive months (8 weekly sessions).

ELIGIBILITY:
Inclusion Criteria:

* TBI of at least mild severity using criteria related to disturbance of consciousness (VHA TBI Comprehensive Evaluation screening tool).
* Obtained informed consent.
* Males or females of working age, between the ages of 18 and 55.
* Medically stable with physician approval to participate
* Ability to comprehend and communicate in English at a 6th grade level
* Executive dysfunction as identified by Frontal Systems Rating Scale (FrSBe) and/or other study assessments

Exclusion Criteria:

* Unable to provide informed consent and no proxy available.
* Severe impairment of language or day- to-day memory that would preclude participation in a verbally-based therapy.
* Life expectancy of less than 36 months.
* Severe multiple trauma (as judged by the attending physicians and/or investigators that is too severe to participate in this study) such as:

  * severe burns
  * serious organ damage
  * amputations
  * multiple fractures
* History of substance abuse severe enough to cause neurologic damage, pre-morbid history of neurologic disease (e.g., stroke).
* Prior history of known bipolar disorder or schizophrenia or severe psychiatric illness as determined by medical history.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 91 (Actual)
Dates: Start 2014-03-12 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2018-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Scholten, MD, Principal Investigator — DCVAMC
Locations (1):
- Washington DC VA Medical Center, Washington, DC, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Libin AV, Scholten J, Schladen MM, Danford E, Shara N, Penk W, Grafman J, Resnik L, Bruner D, Cichon S, Philmon M, Tsai B, Blackman M, Dromerick A. Executive functioning in TBI from rehabilitation to social reintegration: COMPASS (goal,) a randomized controlled trial (grant: 1I01RX000637-01A3 by the VA ORD RR&D, 2013-2016). Mil Med Res. 2015 Nov 30;2:32. doi: 10.1186/s40779-015-0061-2. eCollection 2015. PMID 26664736
- [Result] Libin AV, Schladen MM, Danford E, Cichon S, Bruner D, Scholten J, Llorente M, Zapata S, Dromerick AW, Blackman MR, Magruder KM. Perspectives of veterans with mild traumatic brain injury on community reintegration: Making sense of unplanned separation from service. Am J Orthopsychiatry. 2017;87(2):129-138. doi: 10.1037/ort0000253. PMID 28206800
- See also: Libin, Scholten et al. Perspectives of veterans with mild traumatic brain injury on community reintegration — https://www.ncbi.nlm.nih.gov/pubmed/28206800
- See also: Libin, Scholten et al. Executive functioning in TBI from rehabilitation to social reintegration — https://www.ncbi.nlm.nih.gov/pubmed/26664736

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1: Experimental: The COMPASS (Community Participation through Self-Efficacy Skills Development) program aims at developing and testing a novel patient-centered intervention framework that can be utilized as a platform for VA community re-integration comparative effectiveness research.
  Experimental - COMPASS: Controlled randomized clinical trial. Fifty-five participants in the intervention group will receive eight goal self-management sessions over a period of approximately ten weeks.
- Arm 1: Control: Fifty-five participants in the supported discharge, or control, group will not receive the intervention, but will receive phone calls to answer a short questionnaire and check in on their status.
  Control
  Control - COMPASS: Increased hours of patient-provider interactions Group.
Period: Overall Study
Arm/Group | Arm 1: Experimental | Arm 1: Control
Started | 40 | 51
Completed | 27 | 27
Not Completed | 13 | 24
Not completed — Lost to Follow-up | 13 | 24

BASELINE CHARACTERISTICS:
Groups:
- Experimental - COMPASS: The COMPASS (Community Participation through Self-Efficacy Skills Development) program aims at developing and testing a novel patient-centered intervention framework that can be utilized as a platform for VA community re-integration comparative effectiveness research.
  Experimental - COMPASS: Controlled randomized clinical trial. Fifty-five participants in the intervention group will receive eight goal self-management sessions over a period of approximately ten weeks.
- Control - COMMPASS: Fifty-five participants in the supported discharge, or control, group will not receive the intervention, but will receive phone calls to answer a short questionnaire and check in on their status.
  Control
  Control - COMPASS: Increased hours of patient-provider interactions Group.
- Total: Total of all reporting groups
Arm/Group | Experimental - COMPASS | Control - COMMPASS | Total
Number analyzed (Participants) | 27 | 27 | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 27 | 27 | 54
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (8.3) | 39.6 (6.9) | 39.7 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 22 | 23 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 27 | 27 | 54
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 27 | 27 | 54

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Community Reintegration for Injured Service Members at 2 Months
Description: Change from Baseline in Community Reintegration for Injured Service Members (CRIS) at 2 months. The investigators used in the report CRIS subscale - Extent of Participation, CRIS with the score range 28.0-64.0. Higher scores mean a better outcome for the Extent of Participation, Community Reintegration for Injured Service Members (CRIS)
Time Frame: Baseline and 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Experimental | Arm 1: Control
Number analyzed (Participants) | 27 | 27
score on a scale | 40.22 (5.56) | 37.79 (6.04)

2. Primary Outcome: Change From Baseline in Frontal Systems Behavior Scale at 2 Months
Description: Change from Baseline in Frontal Systems Behavior Scale (FrSBe) at 2 months. Minimum value =21, Maximum value=158, Higher score correlates with worse outcome.
Time Frame: Baseline and 2 months
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1: Experimental | Arm 1: Control
Number analyzed (Participants) | 27 | 27
score on a scale | 85.4 (12.2) | 84.3 (13.12)

ADVERSE EVENTS:
Time Frame: 4 years
Description: Veterans were contacted per protocol, both those in the study arm and the control arm. In addition study participants continued to receive clinical care from the Polytrauma team at the Washington DC VA Medical Center where they were routinely assessed for their reported clinical concerns.
  during the study period no adverse events were reported
Arm/Group | Arm 1: Experimental | Arm 1: Control
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/51
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/51
Other Adverse Events (participants affected / at risk) | 0/40 | 0/51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-08-07): https://cdn.clinicaltrials.gov/large-docs/61/NCT01816061/Prot_SAP_000.pdf